CLINICAL TRIAL: NCT01959243
Title: A Multi-Center, Double-Masked, Randomized, Vehicle-Controlled, Parallel-Group Study Evaluating the Safety of Brimonidine Tartrate Ophthalmic Solution 0.025% Used Four Times Daily in a Population of Pediatric, Adult, and Geriatric Subjects
Brief Title: Safety of Brimonidine Tartrate Ophthalmic Solution in a Population of Pediatric, Adult, and Geriatric Participants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 862
Record Dates: First submitted 2013-10-08; First posted 2013-10-09 (Estimated); Results first posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-09

CONDITIONS: Hyperemia
Keywords: Ocular redness
MeSH Terms: conditions — Hyperemia | interventions — Brimonidine Tartrate; Fluorescein

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brimonidine Tartrate (Experimental): Participants will apply 1 drop of brimonidine tartrate ophthalmic solution 0.025% into each eye 4 times daily for up to 4 consecutive weeks.
  Interventions: Drug: Brimonidine Tartrate; Drug: Sodium Fluorescein; Drug: Fluorescein Sodium and Benoximate Hydrocholoride Ophthalmic Solution USP
- Brimonidine Tartrate Vehicle (Placebo Comparator): Participants will apply 1 drop of the vehicle of brimonidine tartrate ophthalmic solution into each eye 4 times daily for up to 4 consecutive weeks.
  Interventions: Drug: Vehicle; Drug: Sodium Fluorescein; Drug: Fluorescein Sodium and Benoximate Hydrocholoride Ophthalmic Solution USP

INTERVENTIONS:
Drug: Brimonidine Tartrate — Ophthalmic solution to be applied as directed.
  Arms: Brimonidine Tartrate
Drug: Vehicle — Ophthalmic solution to be applied as directed.
  Arms: Brimonidine Tartrate Vehicle
Drug: Sodium Fluorescein — For use as needed during the study for evaluating corneal damage.
Drug: Fluorescein Sodium and Benoximate Hydrocholoride Ophthalmic Solution USP — For use as needed during the study for intraocular pressure and dilated ophthalmoscopy.

SUMMARY:
To compare the safety and tolerability of brimonidine tartrate ophthalmic solution 0.025% versus its vehicle in a population of pediatric, adult, and geriatric participants. At least 51% of participants will be 40 years of age or older.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 5 years of age at Baseline (Visit 1) of either sex and any race or ethnicity;
* Have ocular health within normal limits, including a calculated best-corrected (if necessary) visual acuity of 0.3 logarithm of the minimum angle of resolution (logMAR) or better in each eye, as measured using an Early Treatment of Diabetic Retinopathy Study (ETDRS) chart.

Exclusion Criteria:

* Have any ocular/systemic health problems
* Use of any disallowed medications during the period indicated prior to Baseline (Visit 1) and for the duration of the study.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 507 (Actual)
Dates: Start 2014-02-22 (Actual); Primary Completion 2014-04-23 (Actual); Study Completion 2014-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heleen DeCory, Study Director — Bausch & Lomb Incorporated
Locations (4):
- United States (4):
  - Bausch Site 3, Phoenix, Arizona
  - Bausch Site 4, Havre de Grace, Maryland
  - Bausch Site 1, Andover, Massachusetts
  - Bausch Site 2, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized in a 2:1 ratio to receive brimonidine tartrate ophthalmic solution or the vehicle of brimonidine tartrate ophthalmic solution, respectively.
Groups:
- Brimonidine Tartrate: Participants applied 1 drop of brimonidine tartrate ophthalmic solution 0.025% into each eye 4 times daily for up to 4 consecutive weeks.
- Brimonidine Tartrate Vehicle: Participants applied 1 drop of the vehicle of brimonidine tartrate ophthalmic solution into each eye 4 times daily for up to 4 consecutive weeks.
Period: Overall Study
Arm/Group | Brimonidine Tartrate | Brimonidine Tartrate Vehicle
Started | 337 | 170
Received at Least 1 Dose of Study Drug | 337 | 170
Completed | 324 | 166
Not Completed | 13 | 4
Not completed — Investigator Decision | 3 | 0
Not completed — Adverse Event | 5 | 2
Not completed — Administrative reasons | 2 | 1
Not completed — Lost to Follow-up | 3 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug (Safety Population).
Groups:
- Total: Total of all reporting groups
Arm/Group | Brimonidine Tartrate | Brimonidine Tartrate Vehicle | Total
Number analyzed (Participants) | 337 | 170 | 507
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (17.13) | 41.0 (17.68) | 40.8 (17.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 200 | 100 | 300
  Male | 137 | 70 | 207

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: TEAE is defined as any untoward medical occurrence or undesirable event(s) that begins or worsens following administration of the study drug, whether or not considered related to the treatment by the Investigator. A TEAE is considered serious if, in the view of the Investigator or Sponsor, it results in any of the following outcomes: death, a life-threatening TEAE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, an important medical event that jeopardized the participant and required medical intervention, or sight-threatening (possibly resulting in persistent or significant loss of vision). A summary of other non-serious adverse events (AEs) and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to Day 29
Population: All randomized participants who received at least 1 dose of study drug (Safety Population).
Measure: Count of Participants; unit: Participants
Arm/Group | Brimonidine Tartrate | Brimonidine Tartrate Vehicle
Number analyzed (Participants) | 337 | 170
Participants
  Participants with at Least 1 TEAE | 66 | 38
  Participants with at Least 1 Ocular TEAE | 44 | 25
  Participants with at least 1 Non-Ocular TEAE | 23 | 16
  Participants with at least 1 Serious TEAE | 2 | 0
  Participants Discontinued from Study due to TEAEs | 5 | 2

2. Secondary Outcome: Drop Comfort Assessment as Assessed by the Participant
Description: Drop comfort assessment (0-10 unit scale in which a score of 0 denotes "very comfortable" and 10 is "very uncomfortable") was performed by the participant. Participant's average score across eyes at each time point were used for analysis.
Time Frame: At dose installation, 30 seconds postdose installation, and 1 minute postdose installation on Day 1
Population: All randomized participants who received at least 1 dose of study drug (Safety Population).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Brimonidine Tartrate | Brimonidine Tartrate Vehicle
Number analyzed (Participants) | 337 | 170
units on a scale
  Upon Dose Installation | 0.4 (0.90) | 0.4 (0.77)
  30 Seconds Postdose Installation | 0.4 (0.90) | 0.3 (0.85)
  1 Minute Postdose Installation | 0.4 (0.83) | 0.4 (0.83)

3. Secondary Outcome: Number of Participants Who Were Fully Alert as Assessed by the Investigator on Days 1, 8, 15, and 29
Description: An alertness evaluation was performed by the Investigator asking the participant and/or participant's parent/legal guardian (pediatric participants only) a few questions based on the previous week. Using those answers, along with his/her clinical opinion, the Investigator made an assessment of the participant's level of alertness using the following 6-point scale: fully alert, alert, lethargy, obtunded, stupor, or coma.
Time Frame: Predose installation on Day 1 and 90-180 minutes postdose installation on Days 1, 8, 15, and 29
Population: All randomized participants who received at least 1 dose of study drug (Safety Population) with evaluable alertness data.
Measure: Count of Participants; unit: Participants
Arm/Group | Brimonidine Tartrate | Brimonidine Tartrate Vehicle
Number analyzed (Participants) | 337 | 170
Participants
  Predose Installation on Day 1 | 337 | 170
  Postdose Installation on Day 1: number analyzed (Participants) | 336 | 169
  Postdose Installation on Day 1 | 336 | 169
  Postdose Installation on Day 8: number analyzed (Participants) | 326 | 167
  Postdose Installation on Day 8 | 326 | 167
  Postdose Installation on Day 15: number analyzed (Participants) | 326 | 166
  Postdose Installation on Day 15 | 326 | 166
  Postdose Installation on Day 29: number analyzed (Participants) | 323 | 164
  Postdose Installation on Day 29 | 323 | 164

ADVERSE EVENTS:
Time Frame: Baseline up to Day 29
Description: All randomized participants who received at least 1 dose of study drug (Safety Population).
Arm/Group | Brimonidine Tartrate | Brimonidine Tartrate Vehicle
Serious Adverse Events (participants affected / at risk) | 2/337 | 0/170
Other Adverse Events (participants affected / at risk) | 27/337 | 14/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brimonidine Tartrate (N=337) | Brimonidine Tartrate Vehicle (N=170)
Gastroenteritis (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brimonidine Tartrate (N=337) | Brimonidine Tartrate Vehicle (N=170)
Visual Acuity Reduced (Eye disorders) | 16 | 9
Conjunctival Hyperaemia (Eye disorders) | 11 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact Sponsor directly for additional information.